CLINICAL TRIAL: NCT01869023
Title: Phase II Study of Six Hours, Low Dose Gemcitabine Plus Cisplatin in the Treatment for Advanced Pleural Mesothelioma.
Brief Title: Phase II Study of Six Hours Low Dose Gemcitabine Plus Cisplatin in the Treatment for Advanced Pleural Mesothelioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez MD, Chief of Thoracic Oncology Department, Instituto Nacional de Cancerologia de Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCANOGAR2012-JA3
Record Dates: First submitted 2012-04-18; First posted 2013-06-05 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Advanced Malignant Pleural Mesothelioma
Keywords: Advanced Malignant Pleural Mesothelioma; Gemcitabine and cisplatin; Gemcitabine continuous infusion
MeSH Terms: interventions — Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 6 h infusion Gemcitabine and Cisplatin (Other): Gemcitabine 250 mg/m2 Cisplatin 30 mg/m2
  Interventions: Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Gemcitabine — Combination of Gemcitabine 250 mg/m2 in six hour infusion with cisplatin 35 mg/m2 administered day 1 and 8, for six cycles.
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin 35 mg/m2SC applied on day 1 of 3 weeks cycles
  Other Names: Platinol

SUMMARY:
Malignant pleural mesothelioma (MPM) is a rare disease, but with a very high mortality. MPM is frequently found in advanced stages. The standard treatment in advanced pleural mesothelioma is cisplatin-based chemotherapy combined with pemetrexed/raltitrexed (phase III studies showed its benefit in response and overall survival compared with cisplatin alone). There are other active drugs such as liposomal doxorubicin and gemcitabine. Unfortunately, cost is an important factor to consider in our population and standard treatments are very expensive. Gemcitabine 250 mg infused over 6 hrs in combination with cisplatin, compared to the standard administration of gemcitabine 1250 mg infusion of 30 minutes in NSCLC, combined with cisplatin showed 75 mg shown in a study to be equally effective in treating cancer non-small cell lung. A phase II study using this strategy for advanced MPM has shown promising results. Gemcitabine administered in low dose in a six hour infusion may reduce cost of treatment without altering the effectiveness.

Primary Objective.

-Evaluate the response of treatment with gemcitabine at a dose of 250 mg/m2SC in 6-hour infusion combined with cisplatin in patients with unresectable malignant mesothelioma.

Secondary objectives.

* Evaluate toxicity of the combination of gemcitabine at a dose of 250 mg/m2 infused over 6 hours in with cisplatin in patients with unresectable malignant mesothelioma.
* Evaluate the progression free survival (PFS) and overall survival (OS) in patients with unresectable MM treated with this combination.

Hypothesis:

Combination therapy of gemcitabine at a dose of 250 mg/m2 infusion of 6 hrs applied on day 1 and 8 combined with cisplatin 35 mg/m2SC applied on day 1 of 3 weeks cycles is a treatment that provides similar results in responses when compared with previous studies with the same combination therapy, but with a conventional administration (gemcitabine 1,250 mg in 30 minutes on days 1, 8 and 15).

DETAILED DESCRIPTION:
Malignant pleural mesothelioma is a rare disease, but with a high mortality. It usually develops in people who were exposed to asbestos, with a latency period ranging from 20 to 40 years. Most of these patients present with advanced disease, which are considered unresectable and combination chemotherapy is the treatment of choice. Currently the standard treatment is the combination of pemetrexed with cispaltin, this treatment showed benefit in overall survival and overall response rate in comparison with the treatment with cisplatin alone. This standard chemotherapy in our country is difficult to access due to the costs of the treatment and the poor economic situation of most of our patients. That's why determining the effectiveness of other treatment options that have shown activity in this disease that are less expensive, is of vital importance in our country. Phase I studies of gemcitabine showed that the maximum tolerated dose varies with time of infusion, 250 mg/m2 is the maximum tolerated dose when the infusion is carried out in 6 hours, as opposed to 1250 mg/m2 when gemcitabine is administered in a conventional manner . A phase III study in NSCLC, which compared the administration of gemcitabine infusion of 250 mg/m2 in 6 hours versus conventional administration of 1,250 mg/m2 in 30 minutes showed that both treatments were similar in efficacy and toxicity. The same group conducted a phase II study in unresectable malignant pleural mesothelioma that was published recently with promising results. That is why we decided to conduct a phase II study in patients with unresectable malignant pleural mesothelioma with the idea of validating the results previously obtained and to study factors and associated with resistance to chemotherapy as ERCC1, RPM1, thymidylate synthase.

ELIGIBILITY:
Inclusion Criteria:

* Histologic Diagnosis of Pleural Mesothelioma
* Multidisciplinary assessment and considered not candidate for resection.
* Karnofsky > = 70 or ECOG < 2
* Adequate Hematologic, renal and hepatic function.

Exclusion Criteria:

* Superior vena cava syndrome, severe bone pain or CNS metastasis
* Not candidate for chemotherapy (Poor functional status: ECOG > 2)
* The patient refuses to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2010-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate adverse effects to 250 mg/m2 infusion gemcitabine | 2 years

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD, Principal Investigator — Instituto de Cancerología
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Arrieta O, Lopez-Macias D, Mendoza-Garcia VO, Bacon-Fonseca L, Munoz-Montano W, Macedo-Perez EO, Muniz-Hernandez S, Blake-Cerda M, Corona-Cruz JF. A phase II trial of prolonged, continuous infusion of low-dose gemcitabine plus cisplatin in patients with advanced malignant pleural mesothelioma. Cancer Chemother Pharmacol. 2014 May;73(5):975-82. doi: 10.1007/s00280-014-2429-5. Epub 2014 Apr 1. PMID 24687408